CLINICAL TRIAL: NCT06372262
Title: Effect of 2000-meter Rowing Test on Parameters of Intestinal Integrity in Elite Rowers During Competitive Phase
Acronym: Rowers
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Rowers2022
Record Dates: First submitted 2024-03-19; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2022-06

CONDITIONS: Endothelial Dysfunction
Keywords: endotoxin; gastrointestinal symptoms; gut permeability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ergometer test — 2000meter rowing ergometer test

SUMMARY:
The study aimed to check the 2000m ergometer test on markers of gut permeability in the competitive phase of rowers. 18 members of the Polish rowing team took part in the study.

DETAILED DESCRIPTION:
The phenomenon of epithelial wall leakage has been the subject of investigations within athletic domains such as running and cycling. Nevertheless, there exists an insufficiency of understanding regarding gut permeability in alternative disciplines, such as rowing, particularly following the completion of a standard competitive distance of 2000 meters. Hence, the principal objective of our study was to assess gut permeability after completing a 2000-meter rowing test. The study was performed at the beginning of a competitive training phase. Eighteen elite Polish Rowing Team rowers participated in the study after applying the inclusion/exclusion criteria. The participants performed a 2000-meter ergometer test. Blood samples were taken before the test, after exercise, and after 1-hour of restitution. Parameters, such as I-FABP, LPS, LBP, and zonulin, were determined using appropriate biochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* minimum five years of training,
* five training sessions per week minimum,
* total training time minimum of 240 minutes,
* membership in the Polish Rowing Team,
* finishing the 2000-meter ergometer test.

Exclusion Criteria:

* antibiotic therapy within the last three months,
* probiotics and prebiotics within the last three months,
* dietary regime,
* gastrointestinal diseases.

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male rowers age 18 - 22 years.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
I-FABP (intestinal fatty acid binding protein)to measure epithelial wall injury | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  I-FABP concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
zonulin to measure tight junction leakage | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  zonulin concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
LBP (lipopolysaccharide binding protein) to measure endotoxin | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  LBP concentration measured in blood [ug/ml] using commercially available enzyme-linked immunosorbent assays
LPS (lipopolysaccharide) to measure endotoxin | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 1-hour recovery period
  LPS concentration measured in blood [EU/Ll] using commercially available enzyme-linked immunosorbent assays
Lactic acid to measure fatigue after the race | Blood samples was taken from earlobe at two-time points: before each stress test (after overnight fasting), one minute after the end of the test.
  Lactate concentration measured in capillary blood from earlobe [mmol/L] using a commercially available kit (Diaglobal, Berlin, Germany)

SECONDARY OUTCOMES:
energy | day before test
  energy [kcal ]of food intake measured by 24h dietary recall
fiber intake | day before test
  fiber [g] intake day before the test measured by 24h dietary recall
protein | day before test
  protein [g] intake day before the test measured by 24h dietary recall
carbohydrate | day before test
  carbohydrate [g] intake day before the test measured by 24h dietary recall
body mass | in the morning before the test
  Body mass [kg] measured by electronic scale to the nearest 0,05 kg (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Body composition - water | in the morning before the test
  % of body water measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Body composition - fat | in the morning before the test
  % of body fat measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Lean body mass | in the morning before the test
  Lean body mass [kg] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejnborn, proffessor, Study Director — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No